CLINICAL TRIAL: NCT00052273
Title: A Phase I Dose Escalation Study With Oral LY317615 in Combination With Capecitabine in Advanced Cancer Patients
Brief Title: LY317615 Plus Capecitabine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000258138; UCLA-0206061; LILLY-H6Q-MC-JCAH; NCI-G02-2132
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Adult; Solid Tumor
Keywords: unspecified adult solid tumor; protocol specific
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Drug: enzastaurin hydrochloride

SUMMARY:
RATIONALE: LY317615 may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth and by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining LY317615 with capecitabine may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining LY317615 with capecitabine in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and the recommended phase II dose of LY317615 and capecitabine in patients with advanced solid tumors.
* Determine the safety profile of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine, preliminarily, the antitumor activity of this regimen in these patients.
* Determine the effects of LY317615 on potential angiogenic surrogate markers in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral LY317615 daily on days 1-14 (course 1 only). Beginning with course 2, patients receive oral LY317615 daily on days 1-21 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of LY317615 and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the recommended phase II dose.

Patients are followed at 30 days after the last dose of study drug.

PROJECTED ACCRUAL: A total of 12-36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor that is refractory to standard therapy or for which no standard therapy exists
* Measurable or evaluable disease
* 18 and over
* ECOG 0-2
* Hematopoietic

  * Absolute neutrophil count at least 1,500/mm^3
  * Platelet count at least 100,000/mm^3
  * Hemoglobin at least 9 g/dL (erythrocyte transfusions allowed)
* Hepatic

  * Bilirubin no greater than 1.5 times upper limit of normal (ULN)
  * ALT and AST no greater than 2.5 times ULN (5 times ULN if liver metastases present)
* Renal

  * Creatinine clearance at least 50 mL/min
  * Potassium at least 3.4 mEq/L
  * Calcium at least 8.4 mg/dL
  * Magnesium at least 1.2 mEq/L
* Cardiovascular

  * QTc interval no greater than 450 msec in males
  * QTc interval no greater than 470 msec in females
  * No other electrocardiogram abnormalities
* Able to swallow capsules
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3-6 months after study
* Endocrine therapy

  * At least 4 weeks since prior anticancer hormonal therapy
  * At least 6 weeks since prior bicalutamide
  * At least 4 weeks since prior flutamide or nilutamide
  * Concurrent luteinizing hormone-releasing hormone analog therapy (e.g., leuprolide or goserelin) allowed for patients with prostate cancer if started before study entry
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin).
* Radiotherapy

  * At least 4 weeks since prior radiotherapy
  * At least 2 weeks since prior palliative radiotherapy
  * Recovered from prior therapy
* Other

  * At least 4 weeks since prior investigational anticancer therapy
  * At least 4 weeks since other prior anticancer therapy
  * At least 30 days since prior experimental drugs

Exclusion Criteria:

* known untreated or symptomatic CNS metastases
* concurrent hematologic malignancies
* gastrointestinal disorder that would interfere with oral drug absorption
* serious concurrent systemic disorder
* compliance issues that would preclude study
* geographical conditions that would preclude study
* active infection
* prior hypersensitivity to any component of study drugs
* pregnant or nursing
* concurrent immunotherapy
* concurrent routine filgrastim (G-CSF)
* other concurrent chemotherapy
* other concurrent hormonal therapy
* concurrent radiotherapy (including palliative therapy)
* other concurrent experimental medications
* other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-12; Primary Completion 2004-11 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Britten, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States